CLINICAL TRIAL: NCT01448213
Title: Comparison Of Two Corticosteroid Dosing Regimens For Prevention Of Corneal Transplant Rejection Episodes After Descemet's Membrane Endothelial Keratoplasty
Brief Title: Comparison of Two Steroid Regimens to Prevent Transplant Rejection After Corneal Transplant (DMEK)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Price Vision Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-0329
Record Dates: First submitted 2011-10-04; First posted 2011-10-07 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Fuchs' Dystrophy; Bullous Keratopathy
Keywords: DMEK; Rejection; Corticosteroid
MeSH Terms: conditions — Corneal dystrophy, Fuchs' endothelial, 1; Rejection, Psychology | interventions — prednisolone acetate; Fluorometholone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluorometholone 0.1% Solution (Active Comparator): Subjects assigned to Treatment Regimen B will instill 1 drop of prednisolone acetate 1% four times a day in the transplant eye for one month. Then they will instill one drop of fluorometholone four times a day in the transplant eye for 2 months, then 3 times a day for 1 month, then twice a day for 1 month, then once a day until the subject exits the study.
  Interventions: Drug: Fluorometholone
- Prednisolone acetate 1% Solution (Active Comparator): Subjects assigned to Treatment Regimen A will instill 1 drop of prednisolone acetate 1% four times a day in the transplant eye for 3 months, then 3 times a day for one month, then twice a day for one month, then once a day until the subject exits the study.
  Interventions: Drug: Prednisolone acetate

INTERVENTIONS:
Drug: Prednisolone acetate — Subjects assigned to Treatment Regimen A will instill 1 drop of prednisolone acetate 1% four times a day in the transplant eye for 3 months, then 3 times a day for one month, then twice a day for one month, then once a day until the subject exits the study.
  Arms: Prednisolone acetate 1% Solution
Drug: Fluorometholone — Subjects assigned to Treatment Regimen B will instill 1 drop of prednisolone acetate 1% four times a day in the transplant eye for one month. Then they will instill one drop of fluorometholone four times a day in the transplant eye for 2 months, then 3 times a day for 1 month, then twice a day for 1 month, then once a day until the subject exits the study.
  Arms: Fluorometholone 0.1% Solution

SUMMARY:
The purpose of this study is to compare two different commonly used steroid dosing regimens after Descemet's membrane endothelial keratoplasty (DMEK) transplant surgery. The investigators hope to determine if one is more effective at preventing rejection or if both are equally effective.

DETAILED DESCRIPTION:
Graft rejection is one of the leading causes of cornea transplant failure. To help prevent rejection, corticosteroid eye drops are used after transplant surgery. The steroid eye drop dosing regimen varies from surgeon to surgeon, because no studies have been done to determine the optimum dosing regimen.

ELIGIBILITY:
INCLUSION CRITERIA: The following are requirements for inclusion in the study:

* Male or female patient, at least 18 years of age, who is a candidate for DMEK due to corneal endothelial dysfunction or who has undergone DMEK within the last 7 weeks
* Patient is able and willing to administer eye drops.
* Patient is able to comprehend and has signed the Informed Consent form.
* Patient is likely to complete the entire one-year course of the study.
* Patient has best corrected visual acuity (BCVA) of at least 20/200 in the fellow eye.
* Corneal neovascularization will not be judged as an exclusion criteria for the study

EXCLUSION CRITERIA: The following are exclusion criteria for patients in this study:

* A patient with a previous failed graft in the study eye with a history of a prior rejection episode
* A patient exhibiting any intraocular inflammation
* A patient with a known sensitivity to any of the ingredients in the study medications
* A patient who has a condition (i.e., UNCONTROLLED systemic disease) or is in a situation which in the investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study
* A patient with abnormal eyelid function
* A patient that is exhibiting active corneal ulceration, keratitis, or conjunctivitis, or who has a history of herpetic keratitis
* A patient with the presence of any ocular disease that would interfere with the evaluation of the study treatment
* A patient with a history of non-compliance with using prescribed medication
* A patient who is concurrently involved in or participated in another clinical trial within 30 days prior to enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, MD, Principal Investigator — Price Vision Group; Friedrich Kruse, MD, Principal Investigator — University of Erlangen, Germany
Locations (2):
- Price Vision Group, Indianapolis, Indiana, United States
- University of Erlangen, Erlangen, Germany

REFERENCES:
- [Result] Price MO, Price FW Jr, Kruse FE, Bachmann BO, Tourtas T. Randomized comparison of topical prednisolone acetate 1% versus fluorometholone 0.1% in the first year after descemet membrane endothelial keratoplasty. Cornea. 2014 Sep;33(9):880-6. doi: 10.1097/ICO.0000000000000206. PMID 25062336
- See also: Price Vision Group Website — http://www.pricevisiongroup.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluorometholone 0.1% Solution | Prednisolone Acetate 1% Solution
Started | 130 | 134
Completed | 113 | 112
Not Completed | 17 | 22
Not completed — Lost to Follow-up | 12 | 10
Not completed — Adverse Event | 4 | 10
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data are reported in units of "eyes" as this presentation is most relevant to the assessments presented in the Outcome Measures module.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluorometholone 0.1% Solution | Prednisolone Acetate 1% Solution | Total
Number analyzed (Participants) | 161 | 164 | 325
Age, Continuous [Median (Full Range); unit: years] | 69 [35 to 91] | 67 [42 to 94] | 68 [35 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 105 | 212
  Male | 54 | 59 | 113

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With Immunologic Graft Rejection Episodes
Time Frame: Within 1 year
Measure: Number; unit: eyes
Units Other Than Participants: Number of Eyes
Arm/Group | Fluorometholone 0.1% Solution | Prednisolone Acetate 1% Solution
Number analyzed (Participants) | 130 | 134
Number analyzed (Number of Eyes) | 161 | 164
eyes | 2 | 0
Statistical Analysis 1: Comparison: Fluorometholone 0.1% Solution vs Prednisolone Acetate 1% Solution; Test type: Superiority or Other; p = 0.17, Log Rank

2. Secondary Outcome: Number of Eyes With Intraocular Pressure (IOP) Elevation
Description: Absolute IOP greater than or equal to 24 mm Hg or a relative increase of 10 mm Hg over the baseline preoperative reading.
Time Frame: one day, two days, one week, one month, 3 months, 6 months and 12 months after DMEK
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Fluorometholone 0.1% Solution | Prednisolone Acetate 1% Solution
Number analyzed (Participants) | 130 | 134
Number analyzed (eyes) | 161 | 164
eyes | 9 | 32
Statistical Analysis 1: Comparison: Fluorometholone 0.1% Solution vs Prednisolone Acetate 1% Solution; Test type: Superiority or Other; p = 0.0005, Log Rank

ADVERSE EVENTS:
Arm/Group | Fluorometholone 0.1% Solution | Prednisolone Acetate 1% Solution
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/134
Other Adverse Events (participants affected / at risk) | 0/130 | 13/134
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluorometholone 0.1% Solution (N=130) | Prednisolone Acetate 1% Solution (N=134)
Intraocular pressure control problem requiring discontinuation of study drug (Eye disorders) | 0 (0) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No